CLINICAL TRIAL: NCT03645681
Title: A Study to Evaluate the Safety and Effectiveness of the InnAVasc Arteriovenous Graft for Hemodialysis Access in Patients With End-Stage Renal Disease
Brief Title: Evaluating the Safety and Effectiveness of the InnAVasc Graft for Dialysis Access in Patients With Kidney Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Concerns around a high rate of thrombosis associated with kinking between the pod and the non-ringed graft.
Sponsor: W.L.Gore & Associates (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-1001; 2R44DK108488-02 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-05

CONDITIONS: Kidney Failure, Chronic; Renal Dialysis
Keywords: Vascular Access; Hemodialysis Access; End Stage Renal Disease; Kidney Failure; Hemodialysis; Arteriovenous Graft; AVG; Cannulation; Quick Sealing dialysis graft
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be implanted with an InnAVasc AVG in the forearm or upper arm using standard vascular surgical techniques. There are two model versions of the InnAVasc Graft. The looped model and the straight model. The graft will be placed in a "straight" (soft "C") configuration in the upper arm, or looped configuration in the forearm (forearm loop) or upper arm (axillary loop).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- InnAVasc AVG treatment (Experimental): Patients will be surgically implanted with an InnAVasc AVG in the forearm or upper arm using standard vascular surgical techniques. The graft will be placed in a "straight" (soft "C") configuration in the upper arm, or looped configuration in the forearm (forearm loop) or upper arm (axillary loop).
  Interventions: Device: InnAVasc arteriovenous graft surgical implant

INTERVENTIONS:
Device: InnAVasc arteriovenous graft surgical implant — An InnAVasc AVG will be surgically implanted into the upper arm or forearm of enrolled participants

SUMMARY:
The CSP-1001 study will evaluate the safety and effectiveness of the InnAVasc arteriovenous graft (AVG) when implanted in and used for hemodialysis in participants suffering from end stage renal failure (ESRD). The InnAVasc AVG is implanted and used similar to other standard of care dialysis grafts currently on the market. However, the InnAVasc AVG has been uniquely designed to potentially allow for immediate needle access (same day as implant surgery as opposed to 2-4 weeks of waiting), to potentially reduce excessive bleeding from the graft after dialysis, and it may provide protection from improper or missed needle cannulation attempts.

DETAILED DESCRIPTION:
The CSP-1001 study will evaluate the safety and effectiveness of the InnAVasc arteriovenous graft (AVG) when implanted in and used for hemodialysis in participants suffering from end stage renal failure (ESRD). The InnAVasc AVG is implanted and used similar to other standard of care dialysis grafts currently on the market. However, the InnAVasc AVG has been uniquely designed to potentially allow for immediate needle access (same day as implant surgery as opposed to 2-4 weeks of waiting), to potentially reduce excessive bleeding from the graft after dialysis, and it may provide protection from improper or missed needle cannulation attempts.

This clinical investigation is a prospective, multi-center, single arm, non-randomized study. Participants with ESRD who require hemodialysis and are suitable for an AVG for hemodialysis access will be eligible for inclusion in the study. Suitable participants will be implanted with an InnAVasc AVG in the forearm or upper arm using standard vascular surgical techniques. The graft will be placed in a "straight" (soft "C") configuration in the upper arm, or looped configuration in the forearm (forearm loop) or upper arm (axillary loop). Twenty-six (26) participants will be enrolled to be implanted with the InnAVasc AVG from up to 7 investigational sites in the United States.

The primary effectiveness endpoint of secondary graft patency will be assessed at 6 months but the total study duration is 24 months. The primary safety endpoint will include characterization of dialysis graft adverse events over 6 months. It is hypothesized that the InnAVasc AVG will provide a secondary patency rate similar to the current standard of care dialysis access grafts on the market, but will have the potential to reduce needle cannulation-related adverse events and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD who are not, or who are no longer, candidates for creation of an autologous AV fistula and therefore need placement of an AV graft to start or maintain hemodialysis therapy;
* Age 18 to 80 years old, inclusive;
* Suitable anatomy for implantation of upper arm "straight" or looped graft, or forearm looped graft (graft not to cross the bend of the elbow);
* For patients NOT on Coumadin / warfarin, international normalized ratio (INR) ≤1.5;
* Able and willing to give informed consent;
* Anticipated life expectancy of at least 1 year.

Additional inclusion criteria on Day 0 (intraoperative):

* Both vessels have been exposed and are deemed appropriate for implantation implantation (i.e. based on the surgeon's opinion, artery is of adequate size, has adequate pulse to support AV access flow and is safely clampable (i.e. artery has lack of significant calcification); and the vein is of adequate size, free of localized sclerosis, and is free of immediate outflow obstruction).

Exclusion Criteria:

* History or evidence of severe cardiac disease (New York Heart Association [NYHA] Functional Class III or IV), myocardial infarction within 6 months prior to enrollment, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina;
* Diabetes with a hemoglobin A1c (HbA1c) > 10%
* For upper arm straight configuration, antecubital fossa crease to axillary crease distance < 18 cm.
* History or evidence of severe peripheral arterial disease in the extremity selected for implant (i.e. arterial inflow insufficient to support hemodialysis access);
* Known or suspected central vein stenosis or obstruction on the side of planned graft implantation;
* In the opinion of the investigator, baseline hypotension, or history of frequent hypotensive episodes during dialysis that puts the patient at increased risk of graft thrombosis;
* In the opinion of the investigator, uncontrolled hypertension;
* Baseline hemoglobin <8 g/dL;
* Baseline platelet count <100,000 or >500,000 cells/mm3;
* Documented history of stroke within 6 months prior to enrollment;
* Treatment with any investigational drug or device within 30 days prior to enrollment;
* Female patients who are pregnant, intending to become pregnant, nursing or intending to breastfeed during the study (pregnancy test may only be omitted, if patient is post-menopausal or has a documented history of hysterectomy);
* History of cancer with active disease or treatment within the previous year, except for non-invasive basal or squamous cell carcinoma of the skin;
* Immunodeficiency, including documented history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) or patients receiving immunosuppressive therapy for treatment of an acute inflammatory event or autoimmune flare. Chronic immunosuppressive therapy is acceptable;
* Documented or suspected hypercoagulable state;
* Bleeding diathesis, other than that associated with ESRD;
* Documented history of heparin-induced thrombocytopenia (HIT);
* Active local or systemic infection as documented from the medical history or bloodwork / blood culture data. If the infection resolves, the subject must be at least one-week post resolution of that infection before implantation;
* Scheduled renal transplant within 6 months;
* Any other condition which in the judgment of the investigator would preclude adequate evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - California Institute of Renal Research, San Diego, California
  - Michigan Vascular Center, Flint, Michigan
  - Greenwood Leflore Hospital, Greenwood, Mississippi
  - Dialysis Access Institute at the Regional Medical Center, Orangeburg, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Inova Health Care Service, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intraoperative enrollment criteria:
  Both vessels have been exposed and are deemed appropriate for implantation (i.e. based on the surgeon's opinion, artery is of adequate size, has adequate pulse to support AV access flow and is safely clampable (i.e. artery has lack of significant calcification); and the vein is of adequate size, free of localized sclerosis, and is free of immediate outflow obstruction).
Groups:
- InnAVasc AVG Treatment: Treatment with the InnAVasc arteriovenous graft (IG).
Period: Overall Study
Arm/Group | InnAVasc AVG Treatment
Started | 26
Primary Endpoint Analyzed | 12
Completed 24 Month | 3
Not Completed | 23
Entered Long Term Follow Up | 3
Completed (Completed long term follow up to date (Feb 2023)) | 1
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | InnAVasc AVG Treatment
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Secondary Patency of InnAVasc AVG at 6 Months
Description: Secondary patency is defined as the number of patients free from abandonment, including surgical or endovascular interventions designed to reestablish AVG patency at the 6 month timepoint.
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | InnAVasc AVG Treatment
Number analyzed (Participants) | 26
Participants | 7

2. Primary Outcome: Incidence of Adverse Events of Special Interest (AESIs) Through 6 Months
Description: Adverse Events of special interest included:
  Infection of the study device, pseudoaneurysm formation at any point along the access circuit requiring surgical/endovascular intervention, including thrombin injection and compression, bleeding from the study graft requiring surgical or endovascular intervention or ≥2 units blood transfusion, hematoma from the study graft requiring surgical or endovascular intervention, seroma from the study graft requiring surgical or endovascular intervention, thrombosis of the study graft.
Time Frame: through 6 months
Measure: Number; unit: Adverse Events
Arm/Group | InnAVasc AVG Treatment
Number analyzed (Participants) | 26
Adverse Events | 56

ADVERSE EVENTS:
Time Frame: Adverse events are evaluated through study completion of 24 months
Arm/Group | InnAVasc AVG Treatment
All-Cause Mortality (participants affected / at risk) | 3/26
Serious Adverse Events (participants affected / at risk) | 12/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InnAVasc AVG Treatment (N=26)
Hematoma (Vascular disorders) | 1 (1)
Cerebral Infraction with Left Hemiparesis (Nervous system disorders) | 1 (1)
Post Thrombectomy Hematoma (Vascular disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Infection of AV Graft (Infections and infestations) | 3 (4)
Thrombosis of AV Graft (Vascular disorders) | 1 (1)
Bacteremia (Infections and infestations) | 3 (3)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hypotensive Cardiac Event (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Acute Hypoxemic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InnAVasc AVG Treatment (N=26)
Cannulation Complications (Vascular disorders) | 3 (4)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Arteriovenous Graft Site Hematoma (Vascular disorders) | 2 (4)
Arteriovenous graft site infection (Vascular disorders) | 1 (1)
Arteriovenous graft site stenosis (Vascular disorders) | 11 (33)
Arteriovenous graft thrombosis (Vascular disorders) | 20 (47)
Bacteraemia (Infections and infestations) | 2 (2)
Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Eschar (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalaemia (Blood and lymphatic system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1)
Medical device site extravasation (Injury, poisoning and procedural complications) | 2 (2)
Medical device site oedema (Injury, poisoning and procedural complications) | 1 (1)
Medical device site pain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Protein C deficiency (Blood and lymphatic system disorders) | 1 (1)
Seroma (Blood and lymphatic system disorders) | 1 (1)
Steal Syndrome (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vascular Stenosis (Vascular disorders) | 4 (15)
Hypotensive Cardiac Event (Cardiac disorders) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment was terminated before enrollment was completed, and subject attrition rates prevented full analysis of endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03645681/Prot_SAP_ICF_000.pdf